CLINICAL TRIAL: NCT03446794
Title: Registry of Left Atrial Appendage Occlusion With WATCHMAN® Device in Patients With Non-valvular Atrial Fibrillation and End-stage Chronic Kidney Disease on Hemodialysis
Brief Title: Left Atrial Appendage Occlusion With WATCHMAN® Device in Patients With Non-valvular Atrial Fibrillation and End-stage Chronic Kidney Disease on Hemodialysis
Acronym: WATCH-HD
Status: Completed | Type: Observational
Sponsor: Fundación EPIC (Other)
Responsible Party: Sponsor
Other Study IDs: WATCH-HD EPIC-06
Record Dates: First submitted 2018-02-19; First posted 2018-02-27 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Atrial Fibrillation; Heart Diseases; Renal Disease; Bleeding; Arrhythmias, Cardiac; Cardiovascular Diseases
Keywords: Left Atrial Appendage Closure; Watchman device
MeSH Terms: conditions — Atrial Fibrillation; Heart Diseases; Kidney Diseases; Hemorrhage; Arrhythmias, Cardiac; Cardiovascular Diseases | interventions — Safety

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients with NVAF and ESCKD on HD
  Interventions: Other: Non Intervention

INTERVENTIONS:
Other: Non Intervention — To assess the procedural safety and efficacy on stroke and bleeding prevention of LAAC in patients with NVAF and ESCKD on HD
  Other Names: Safety and efficacy

SUMMARY:
Atrial fibrillation (AF) is more common in patients with renal disease compared to the general population an risk increase to as much as 10 times in patients on hemodialysis (HD). Stroke is an important cause of morbidity, mortality and suffering for patients with end-stage chronic kidney disease (ESCKD) on hemodialysis.The risk of bleeding in these patients can be roughly 5-fold higher that without it. Current guidelines recommend the use of oral anticoagulants (AO) to prevent stroke or systemic thromboembolism in high-risk patients with AF. Left atrial appendage occlusion (LAAO) reduces the risk of bleeding while allows thromboembolic stroke prevention. The aim of the study is to assess the procedural safety on stroke and bleeding prevention of LAAC in patients with non-valvular atrial fibrillation (NVAF) and ESCKD on HD.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is more common in patients with renal disease compared to the general population an risk increase to as much as 10 times in patients on hemodialysis (HD). Stroke is an important cause of morbidity, mortality and suffering for patients with end-stage chronic kidney disease (ESCKD) on hemodialysis.The risk of bleeding in these patients can be roughly 5-fold higher that without it. Current guidelines recommend the use of oral anticoagulants (AO) to prevent stroke or systemic thromboembolism in high-risk patients with AF. Left atrial appendage occlusion (LAAO) reduces the risk of bleeding while allows thromboembolic stroke prevention.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years.
* Stage V chronic kidney disease (GFR <15 ml / min) in hemodialysis at the time of left atrial appendage closure.
* History of atrial or valvular fibrillation (paroxysmal, persistent, permanent).
* Less moderate embolic risk (CHA2DS2-VASc ≥2) or active oral anticoagulant therapy due to atrial fibrillation.
* High associated hemorrhagic risk (HASBLED ≥ 3) or a history of major bleeding (BARC> 2).
* The patient has been informed of the characteristics of the study and has provided written informed consent.

Exclusion Criteria:

* Life expectancy < 2 years.
* Indication for OA different from NVAF.
* Severe pericardial effusion.
* Previous percutaneous closure of atrial septal defect.
* Intracardiac thrombus.
* Severe hepatic dysfunction with spontaneous INR (International Normalized Ratio) > 1.5.
* The patient refuses to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients With Non-valvular Atrial Fibrillation and End-stage Chronic Kidney Disease on Hemodialysis .
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2018-03-14 (Actual); Primary Completion 2022-01-07 (Actual); Study Completion 2022-01-07 (Actual)

PRIMARY OUTCOMES:
Composite of all-cause mortality, stroke and bleeding | 24 month
  Composite: Stroke or Transient Ischemic Attack (TIA), Systemic embolism, Major bleeding event (BARC ≥ 2).
  Systemic embolism, Major bleeding event (BARC ≥ 2)

SECONDARY OUTCOMES:
Periprocedural major adverse events | 2 days
  Overall mortality, cardiovascular mortality, ischemic and hemorrhagic stroke, systemic embolization, late device embolization (beyond hospitalization)
Echocardiographic adverse events during follow up | 24 month
  Prevalence of device thrombus
Echocardiographic adverse events during follow up | 24 month
  Prevalence and severity of residual leak

CONTACTS AND LOCATIONS:
Locations (20):
- Spain (20):
  - Hospital de Vinalopó, Torrevieja, Alicante
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - Hospital Costa del Sol, Marbella, Málaga
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Santa Creu y Sant Pau, Barcelona
  - Hospital Universitario Puerta del Mar, Cadiz
  - Hospital Juan Ramón Jiménez Huelva, Huelva
  - Complejo Hospitalario de Jaén, Jaén
  - Hospital Universitario de Gran Canaria Dr. Negrín, Las Palmas de Gran Canaria
  - Hospital Universitario de León, León
  - Hospital Clínico Universitario San Carlos, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital Universitario Virgen de Arrixaca, Murcia
  - Hospital Universitario Central de Asturias, Oviedo
  - Clínica Universitaria de Navarra, Pamplona
  - Hospital Clínico Universitario de Salamanca, Salamanca
  - Hospital Clínico Universitario Santiago de Compostela, Santiago de Compostela
  - Hospital Universitario Virgen de la Macarena, Seville
  - Hospital Universitario Miguel Servet, Zaragoza

REFERENCES:
- [Result] Fabbian F, Catalano C, Lambertini D, Tarroni G, Bordin V, Squerzanti R, Gilli P, Di Landro D, Cavagna R. Clinical characteristics associated to atrial fibrillation in chronic hemodialysis patients. Clin Nephrol. 2000 Sep;54(3):234-9. PMID 11020022
- [Result] Vazquez E, Sanchez-Perales C, Borrego F, Garcia-Cortes MJ, Lozano C, Guzman M, Gil JM, Borrego MJ, Perez V. Influence of atrial fibrillation on the morbido-mortality of patients on hemodialysis. Am Heart J. 2000 Dec;140(6):886-90. doi: 10.1067/mhj.2000.111111. PMID 11099992
- [Result] Wizemann V, Tong L, Satayathum S, Disney A, Akiba T, Fissell RB, Kerr PG, Young EW, Robinson BM. Atrial fibrillation in hemodialysis patients: clinical features and associations with anticoagulant therapy. Kidney Int. 2010 Jun;77(12):1098-106. doi: 10.1038/ki.2009.477. Epub 2010 Jan 6. PMID 20054291
- [Result] Winkelmayer WC, Patrick AR, Liu J, Brookhart MA, Setoguchi S. The increasing prevalence of atrial fibrillation among hemodialysis patients. J Am Soc Nephrol. 2011 Feb;22(2):349-57. doi: 10.1681/ASN.2010050459. Epub 2011 Jan 13. PMID 21233416
- [Result] Providencia R, Marijon E, Boveda S, Barra S, Narayanan K, Le Heuzey JY, Gersh BJ, Goncalves L. Meta-analysis of the influence of chronic kidney disease on the risk of thromboembolism among patients with nonvalvular atrial fibrillation. Am J Cardiol. 2014 Aug 15;114(4):646-53. doi: 10.1016/j.amjcard.2014.05.048. Epub 2014 Jun 6. PMID 25001152
- [Result] Seliger SL, Gillen DL, Longstreth WT Jr, Kestenbaum B, Stehman-Breen CO. Elevated risk of stroke among patients with end-stage renal disease. Kidney Int. 2003 Aug;64(2):603-9. doi: 10.1046/j.1523-1755.2003.00101.x. PMID 12846756
- [Result] Zimmerman D, Sood MM, Rigatto C, Holden RM, Hiremath S, Clase CM. Systematic review and meta-analysis of incidence, prevalence and outcomes of atrial fibrillation in patients on dialysis. Nephrol Dial Transplant. 2012 Oct;27(10):3816-22. doi: 10.1093/ndt/gfs416. PMID 23114904
- [Result] Biggers JA, Remmers AR Jr, Glassford DM, Sarles HE, Lindley JD, Fish JC. The risk of anticoagulation in hemodialysis patients. Nephron. 1977;18(2):109-13. doi: 10.1159/000180784. PMID 854139
- [Result] Holden RM, Harman GJ, Wang M, Holland D, Day AG. Major bleeding in hemodialysis patients. Clin J Am Soc Nephrol. 2008 Jan;3(1):105-10. doi: 10.2215/CJN.01810407. Epub 2007 Nov 14. PMID 18003768
- [Result] Elliott MJ, Zimmerman D, Holden RM. Warfarin anticoagulation in hemodialysis patients: a systematic review of bleeding rates. Am J Kidney Dis. 2007 Sep;50(3):433-40. doi: 10.1053/j.ajkd.2007.06.017. PMID 17720522
- [Result] Clase CM, Holden RM, Sood MM, Rigatto C, Moist LM, Thomson BK, Mann JF, Zimmerman DL. Should patients with advanced chronic kidney disease and atrial fibrillation receive chronic anticoagulation? Nephrol Dial Transplant. 2012 Oct;27(10):3719-24. doi: 10.1093/ndt/gfs346. PMID 23114898
- [Result] Kirchhof P, Benussi S, Kotecha D, Ahlsson A, Atar D, Casadei B, Castella M, Diener HC, Heidbuchel H, Hendriks J, Hindricks G, Manolis AS, Oldgren J, Alexandru Popescu B, Schotten U, Van Putte B, Vardas P. 2016 ESC Guidelines for the Management of Atrial Fibrillation Developed in Collaboration With EACTS. Rev Esp Cardiol (Engl Ed). 2017 Jan;70(1):50. doi: 10.1016/j.rec.2016.11.033. No abstract available. English, Spanish. PMID 28038729
- [Result] Bonde AN, Lip GY, Kamper AL, Hansen PR, Lamberts M, Hommel K, Hansen ML, Gislason GH, Torp-Pedersen C, Olesen JB. Net clinical benefit of antithrombotic therapy in patients with atrial fibrillation and chronic kidney disease: a nationwide observational cohort study. J Am Coll Cardiol. 2014 Dec 16;64(23):2471-82. doi: 10.1016/j.jacc.2014.09.051. PMID 25500231
- [Result] van Latum JC, Koudstaal PJ, Venables GS, van Gijn J, Kappelle LJ, Algra A. Predictors of major vascular events in patients with a transient ischemic attack or minor ischemic stroke and with nonrheumatic atrial fibrillation. European Atrial Fibrillation Trial (EAFT) Study Group. Stroke. 1995 May;26(5):801-6. doi: 10.1161/01.str.26.5.801. PMID 7740570
- [Result] European Atrial Fibrillation Trial Study Group. Optimal oral anticoagulant therapy in patients with nonrheumatic atrial fibrillation and recent cerebral ischemia. N Engl J Med. 1995 Jul 6;333(1):5-10. doi: 10.1056/NEJM199507063330102. PMID 7776995
- [Result] Patients with nonvalvular atrial fibrillation at low risk of stroke during treatment with aspirin: Stroke Prevention in Atrial Fibrillation III Study. The SPAF III Writing Committee for the Stroke Prevention in Atrial Fibrillation Investigators. JAMA. 1998 Apr 22-29;279(16):1273-7. PMID 9565007
- [Result] Lai HM, Aronow WS, Kalen P, Adapa S, Patel K, Goel A, Vinnakota R, Chugh S, Garrick R. Incidence of thromboembolic stroke and of major bleeding in patients with atrial fibrillation and chronic kidney disease treated with and without warfarin. Int J Nephrol Renovasc Dis. 2009;2:33-7. doi: 10.2147/ijnrd.s7781. Epub 2009 Nov 19. PMID 21694919
- [Result] Chan KE, Lazarus JM, Thadhani R, Hakim RM. Warfarin use associates with increased risk for stroke in hemodialysis patients with atrial fibrillation. J Am Soc Nephrol. 2009 Oct;20(10):2223-33. doi: 10.1681/ASN.2009030319. Epub 2009 Aug 27. PMID 19713308
- [Result] Shah M, Avgil Tsadok M, Jackevicius CA, Essebag V, Eisenberg MJ, Rahme E, Humphries KH, Tu JV, Behlouli H, Guo H, Pilote L. Warfarin use and the risk for stroke and bleeding in patients with atrial fibrillation undergoing dialysis. Circulation. 2014 Mar 18;129(11):1196-203. doi: 10.1161/CIRCULATIONAHA.113.004777. Epub 2014 Jan 22. PMID 24452752
- [Result] Genovesi S, Rossi E, Gallieni M, Stella A, Badiali F, Conte F, Pasquali S, Bertoli S, Ondei P, Bonforte G, Pozzi C, Rebora P, Valsecchi MG, Santoro A. Warfarin use, mortality, bleeding and stroke in haemodialysis patients with atrial fibrillation. Nephrol Dial Transplant. 2015 Mar;30(3):491-8. doi: 10.1093/ndt/gfu334. Epub 2014 Oct 28. PMID 25352571
- [Result] Olesen JB, Lip GY, Kamper AL, Hommel K, Kober L, Lane DA, Lindhardsen J, Gislason GH, Torp-Pedersen C. Stroke and bleeding in atrial fibrillation with chronic kidney disease. N Engl J Med. 2012 Aug 16;367(7):625-35. doi: 10.1056/NEJMoa1105594. PMID 22894575
- [Result] Tantisattamo E, Han KH, O'Neill WC. Increased vascular calcification in patients receiving warfarin. Arterioscler Thromb Vasc Biol. 2015 Jan;35(1):237-42. doi: 10.1161/ATVBAHA.114.304392. Epub 2014 Oct 16. PMID 25324574
- [Result] January CT, Wann LS, Alpert JS, Calkins H, Cigarroa JE, Cleveland JC Jr, Conti JB, Ellinor PT, Ezekowitz MD, Field ME, Murray KT, Sacco RL, Stevenson WG, Tchou PJ, Tracy CM, Yancy CW; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2014 AHA/ACC/HRS guideline for the management of patients with atrial fibrillation: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and the Heart Rhythm Society. J Am Coll Cardiol. 2014 Dec 2;64(21):e1-76. doi: 10.1016/j.jacc.2014.03.022. Epub 2014 Mar 28. No abstract available. PMID 24685669
- [Result] Holmes DR Jr, Doshi SK, Kar S, Price MJ, Sanchez JM, Sievert H, Valderrabano M, Reddy VY. Left Atrial Appendage Closure as an Alternative to Warfarin for Stroke Prevention in Atrial Fibrillation: A Patient-Level Meta-Analysis. J Am Coll Cardiol. 2015 Jun 23;65(24):2614-2623. doi: 10.1016/j.jacc.2015.04.025. PMID 26088300
- [Result] Reddy VY, Doshi SK, Sievert H, Buchbinder M, Neuzil P, Huber K, Halperin JL, Holmes D; PROTECT AF Investigators. Percutaneous left atrial appendage closure for stroke prophylaxis in patients with atrial fibrillation: 2.3-Year Follow-up of the PROTECT AF (Watchman Left Atrial Appendage System for Embolic Protection in Patients with Atrial Fibrillation) Trial. Circulation. 2013 Feb 12;127(6):720-9. doi: 10.1161/CIRCULATIONAHA.112.114389. Epub 2013 Jan 16. PMID 23325525
- [Result] Boersma LV, Schmidt B, Betts TR, Sievert H, Tamburino C, Teiger E, Pokushalov E, Kische S, Schmitz T, Stein KM, Bergmann MW; EWOLUTION investigators. Implant success and safety of left atrial appendage closure with the WATCHMAN device: peri-procedural outcomes from the EWOLUTION registry. Eur Heart J. 2016 Aug;37(31):2465-74. doi: 10.1093/eurheartj/ehv730. Epub 2016 Jan 27. PMID 26822918
- [Result] Kefer J, Tzikas A, Freixa X, Shakir S, Gafoor S, Nielsen-Kudsk JE, Berti S, Santoro G, Aminian A, Landmesser U, Nietlispach F, Ibrahim R, Danna PL, Benit E, Budts W, Stammen F, De Potter T, Tichelbacker T, Gloekler S, Kanagaratnam P, Costa M, Cruz-Gonzalez I, Sievert H, Schillinger W, Park JW, Meier B, Omran H. Impact of chronic kidney disease on left atrial appendage occlusion for stroke prevention in patients with atrial fibrillation. Int J Cardiol. 2016 Mar 15;207:335-40. doi: 10.1016/j.ijcard.2016.01.003. Epub 2016 Jan 9. PMID 26820363
- [Result] Meier B, Blaauw Y, Khattab AA, Lewalter T, Sievert H, Tondo C, Glikson M; Document Reviewers. EHRA/EAPCI expert consensus statement on catheter-based left atrial appendage occlusion. Europace. 2014 Oct;16(10):1397-416. doi: 10.1093/europace/euu174. Epub 2014 Aug 29. No abstract available. PMID 25172844